CLINICAL TRIAL: NCT06608251
Title: Association of Plasma Metabolomic Biomarkers with Chronic Ischemic White Matter Injury
Acronym: WML
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20240123-07
Record Dates: First submitted 2024-08-07; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Myelinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: white matter lesion — According to the results of magnetic resonance, they were divided into white matter degeneration group and non-white matter degeneration group

SUMMARY:
The cases were screened according to the inclusion criteria, and after the patients signed the informed consent, the clinical data were collected, the imaging data were evaluated, and blood samples were taken for follow-up measurements. In the early morning of the second day after the patient was enrolled, 5mL of peripheral venous blood was drawn and sent to the neurology laboratory of our hospital for separation, and the detection of plasma metabolomics markers was performed.

DETAILED DESCRIPTION:
In the early morning of the second day after the patient was enrolled, 5mL of peripheral venous blood was drawn and sent to the neurology laboratory of our hospital for separation, and the detection of plasma metabolomics markers was performed.Inluding CRP，Complete blood count，Liver and kidney function indicators，et.

ELIGIBILITY:
Inclusion Criteria：

1. Be older than 45 years old;
2. Patients admitted to the Department of Neurology due to headache, vertigo, anxiety, etc.;
3. There were no symptoms of neurological deficit on physical examination;
4. Able to cooperate with the improvement of brain MRI examination;
5. Sign the informed consent form.

Exclusion Criteria:

1. History of stroke, traumatic brain injury, intracranial tumor, central nervous system infection, active malignant tumor, thyroid disease, autoimmune disease, active or chronic inflammatory disease, severe liver and kidney impairment, etc.;
2. accompanied by neurological deficit symptoms;
3. refusal to participate in the study;
4. Other conditions judged by the investigator to be unsuitable for enrollment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: older than 45 years old and without stoke be able to cooperate with the improvement of brain MRI examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
myelinopathy | 2024.06.01-2027.06.01
  The degree of damage to the white matter of the brain is judged based on the magnetic resonance Fazekas score(1-3), with the higher scores indicating the damage more severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, Doctor, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No